CLINICAL TRIAL: NCT04853472
Title: Menopause Sample Collection
Status: Completed | Type: Observational
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTOCOL-1326
Record Dates: First submitted 2021-04-08; First posted 2021-04-21 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Menopause

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Early Stage Peri-Menopause: Mild cycle irregularity over the last 3-6months (minimum), variation of >6 days in length between consecutive cycles including shortened and longer cycles (but not >60 days in length)
- Late Stage Peri-Menopause: Late stage peri-menopause: Irregular cycles with prolonged periods of amenorrhea >60 days in length (but less than 12 months)
- Post-Menopause: Greater than 12 months since last menstrual period

SUMMARY:
This study will provide daily urine samples from women during early and late stage peri-menopause as well as post-menopause over the course of three calendar months in order to maintain the SPD sample bank.

Urine samples will be received in the clinical laboratory and aliquoted into 2.25ml amounts and stored at -80˚C until required.

Symptom information will also be recorded to determine whether there are any noticeable physiological changes that can be related to stage of the menopause.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Between the ages of 45 and 60 years
* Suspects they are going through or have been through the menopause
* Experiencing cycle irregularities:

  * Early Stage Peri-Menopause: Mild cycle irregularity over the last 3-6months (minimum), variation of >6 days in length between consecutive cycles including shortened and longer cycles (but not >60 days in length)
  * Late stage peri-menopause: Irregular cycles with prolonged periods of amenorrhea >60 days in length (but less than 12 months)
  * Post-Menopause: Greater than 12 months since last menstrual period
* Willing to give informed consent

Exclusion Criteria:

* Use of hormone replacement therapy (HRT)
* Use of hormone contraception
* Hysterectomy and/or oophorectomy
* Pregnant or breast feeding
* Other medical reason for amenorrhea (absence of menstruation)

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female only
Study Population: Healthy female volunteers
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Number of daily urine samples collected from women during various stages of the menopause | 3 months
  Daily urine samples collected

SECONDARY OUTCOMES:
Menopause Symptom Information | 3 months
  Daily recording of experience of a range of menopause symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Raniero Zazzeroni, Study Director — SPD Development Company; Jackie Boxer, Principal Investigator — SPD Development Company
Locations (1):
- SPD Development Company Ltd, Bedford, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD